CLINICAL TRIAL: NCT06985316
Title: An Exploratory Clinical Study Evaluating the Efficacy and Safety of Tunlametinib Combined With Fruquintinib in the Third-line Treatment of Advanced Colorectal Cancer Patients With RAS Mutations.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Huang (Other)
Responsible Party: Sponsor-Investigator, Liu Huang, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202504032
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-03

CONDITIONS: CRC, Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tunlametinib combined with Fruquintinib (Experimental)
  Interventions: Drug: Tunlametinib combined with Fruquintinib

INTERVENTIONS:
Drug: Tunlametinib combined with Fruquintinib — Tunlametinib combined with Fruquintinib

SUMMARY:
This study is a prospective, open-label, single-arm clinical study aimed at evaluating the efficacy and safety of Tunlametinib combined with Fruquintinib in the third-line treatment of advanced colorectal cancer patients with RAS mutations.

ELIGIBILITY:
Inclusion Criteria:

1)18 years old or older, both males and females are allowed; 2)ECOG performance status of 0 or 1; 3)Histologically or cytologically proven advanced colorectal cancer; 4)Previous gene testing results indicate positive RAS mutation; 5)According to RECIST v1.1 assessment, there is at least one measurable lesion; 6)Patients who have previously failed second-line systemic antitumor therapy, and have imaging evidence of disease progression, or who are intolerant to the treatment regimen; patients who have failed front line immunotherapy are allowed to receive cross-line treatment; 7)Expected survival period > 3 months; 8)The main organ functions and bone marrow function are normal, meeting the following requirements:

* Blood routine: Hemoglobin ≥80 g/L (no blood transfusion in the last 14 days); Absolute neutrophil count ≥1.5×10^9/L; Platelet count ≥90×10^9/L;
* Liver function: Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) and Alkaline phosphatase (ALP) ≤2.5×upper limit of normal (ULN); if liver metastasis is present, ALT and AST ≤5×ULN, ALP ≤6×ULN; Total bilirubin ≤1.5×ULN; Albumin ≥30 g/L;
* Kidney function: Serum creatinine ≤1.5×ULN or creatinine clearance calculated by the Cockcroft-Gault formula >60 mL/min;
* Heart function: Echocardiography shows left ventricular ejection fraction (LVEF) ≥55%; ECG QTcF ≤480ms; Creatine kinase (CK) ≤1×ULN, troponin/sensitive troponin ≤1×ULN;
* Coagulation function: International Normalized Ratio (INR) for prothrombin time ≤1.5×ULN; Activated partial thromboplastin time (APTT) ≤1.5×ULN;
* Urinalysis: Urine protein <2; when ≥2, a 24-hour urine protein quantification test should be performed; if the quantification test <1g/24h, they can be included in the group; if urine protein ≥1g/24h, they cannot be included; if urine protein ≥2 without quantification testing, they cannot be included; 9)Able to take oral medication; 10)Women of childbearing age must undergo a pregnancy test (serum or urine) within 14 days prior to enrollment, with negative results, and voluntarily use appropriate contraception during the observation period and for 3 months after the last administration of the study drug; for men, they should be surgically sterilized or agree to use appropriate contraception during the observation period and for 3 months after the last administration of the study drug; 11)Voluntarily participate and sign the informed consent form, expected to have good compliance and be able to cooperate with the study according to the protocol requirements.

Exclusion Criteria:

1. There are contraindications that influence investigators' choices in the use of therapeutic drugs (according to the latest drug instructions).
2. Previously received MEK inhibitors;
3. Within 4 weeks before the first use of the drug, underwent major surgery (excluding biopsies and minor outpatient surgeries, such as the placement of vascular access) or experienced serious trauma;
4. There is the presence of clinically symptomatic third space effusion (such as large pleural effusion or ascites) that cannot be controlled through drainage or other methods;
5. Subjects with symptomatic or untreated brain metastases, leptomeningeal metastases, or spinal cord compression, except for the following conditions: asymptomatic brain metastases (i.e., no progressive central nervous system symptoms caused by brain lesions, no need for corticosteroids or antiepileptic drug treatment, and imaging confirms stability of lesions for ≥4 weeks; for patients who have undergone stereotactic brain radiotherapy or surgical treatment, if there has been no disease progression in the brain for 3 months or more, they can be included;
6. Impaired cardiac function or clinically significant cardiovascular diseases, including any of the following:

   * Acute coronary syndrome occurring within 6 months prior to treatment initiation, including acute myocardial infarction, unstable angina, coronary artery bypass graft surgery, coronary angioplasty, and stent implantation;
   * Symptomatic congestive heart failure (New York Heart Association [NYHA] class ≥ II); evidence of clinically significant arrhythmias and/or conduction abnormalities within 6 months prior to treatment initiation or currently;
   * Poorly controlled hypertension (systolic blood pressure ≥ 150 and/or diastolic blood pressure ≥ 100 mmHg under medication control);
   * Abnormalities in heart valve morphology recorded by echocardiography (≥ grade 2), Note: Patients with grade 1 heart valve morphology abnormalities (such as mild regurgitation/stenosis) are allowed to enroll, but patients with moderate valve thickening are prohibited from enrolling;
   * History of congenital long QT syndrome; or taking medications known to prolong the QT interval and unable to ensure discontinuation during the study.
7. A history of retinal diseases during the past or screening, such as: retinal vein occlusion (RVO), retinal artery occlusion, retinal vasculitis, diabetic retinopathy, hypertensive retinopathy, retinal capillary dilatation (Costs disease), retinal pigment epithelial detachment (RPED), etc.; presence of risk factors for RVO during screening (for example, uncontrolled glaucoma or high intraocular pressure, history of hyperviscosity or hypercoagulable syndromes); retinal diseases such as RPED;
8. Interstitial lung disease or interstitial pneumonia, including patients with clinically significant radiation pneumonia (i.e., those affecting daily activities or requiring intervention treatment);
9. Positive for human immunodeficiency virus (HIV) antibodies, positive for syphilis antibodies (Anti TP), positive for hepatitis C virus (HCV) antibodies and HCV RNA, positive for hepatitis B virus surface antigen (HBsAg) and HBV DNA (positive HBsAg requires further testing for HBV DNA, with HBV DNA ≥ 200 IU/ml or ≥ 10^3 copies/ml);
10. A history of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulators or surgery) within 12 months prior to the start of treatment;
11. It is known that there is a history of acute or chronic pancreatitis within 6 months before the start of treatment;
12. Patients with active gastrointestinal bleeding who require treatment;
13. History of allogeneic bone marrow transplantation or organ transplantation;
14. Within 2 weeks prior to the initial administration of the drug, there are uncontrolled active infectious diseases (e.g., requiring intravenous administration of antibiotics, antifungals, or antiviral medications), or unexplained fever >38.5°C occurs during the screening period / before the first dose of the drug;
15. Incurable electrolyte abnormalities (hypokalemia, hypomagnesemia, hypocalcemia detected through blood biochemical tests);
16. Past or currently existing neuromuscular diseases related to elevated CK (such as inflammatory myopathy, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy, rhabdomyolysis syndrome);
17. Venous or arterial thrombotic events that occurred within the first 6 months prior to the initial use of the drug, such as cerebrovascular accidents (including transient ischemic attacks, intracerebral hemorrhages, cerebral infarctions), deep vein thrombosis, and pulmonary embolism, etc.;
18. Symptoms of grade 3 bleeding as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0) occurred within 4 weeks prior to the first use of the drug;
19. Patients with a history of other malignant tumors in the past 5 years are excluded, except for those who have been completely cured of skin basal cell carcinoma or skin squamous cell carcinoma and cervical carcinoma in situ, and/or any malignant tumor patients who have been cured with no disease or who have been disease-free for at least 5 consecutive years;
20. Those who are allergic to any component of this study drug are known;
21. A clear history of neurological or psychiatric disorders, including epilepsy and dementia;
22. Have received any of the following antitumor treatments prior to the initial study of drug administration (either on the market or in clinical trials): ① Antitumor immunotherapy within 3 weeks; ② Large molecular targeted antitumor therapy such as Bevacizumab within 3 weeks; ③ Chemotherapy or clearly antitumor traditional medicine within 2 weeks; ④ Small molecule targeted antitumor drug treatment within 2 weeks or within 5 half-lives (whichever is longer); ⑤ Subjects who have undergone palliative radiation therapy for bone metastasis within 2 weeks are excluded, but those who have received radiation treatment with an area of ≥30% of the bone marrow within 2 weeks are not allowed to be included;
23. Before studying drug administration, all related toxic reactions from antitumor treatments (such as hair loss, skin pigmentation, grade 2 chemotherapy-related peripheral neurotoxicity, grade 2 toxicities caused by immune checkpoint inhibitors like elevated blood sugar or hypothyroidism, etc.) have not recovered to a level of ≤ grade 1 (as determined by NCI CTCAE v5.0);
24. Patients may be used in conjunction with other anticancer drugs (bisphosphonates for the treatment of bone metastases are acceptable);
25. Uncontrolled comorbidities, including but not limited to severe diabetes (fasting blood glucose > 250 mg/dl or 13.9 mmol/L), or other severe diseases requiring systemic treatment;
26. Vaccination with live vaccines or attenuated vaccines within 4 weeks prior to the first dose (Note: If enrolled, participants must not receive live vaccines during the study treatment period and within 30 days after the last dose of the investigational drug);
27. For premenopausal female subjects (postmenopausal female patients must have been menopausal for at least 12 months to be considered infertile), a positive pregnancy test result; during the study and at least 30 days after the last administration of the study drug, females of childbearing potential who are hoping to become pregnant, breastfeeding, or unwilling to use effective contraceptive methods (including female partners of male subjects);
28. Patients who are undergoing treatment and cannot discontinue intravenous or oral medications that have a prohibitive effect on CYP isoenzymes (strong inducers or strong inhibitors of CYP2C9 and CYP3A4) at least 1 week before starting the study treatment and during the study; patients who are taking medications with a narrow therapeutic window that are metabolized by CYP1A2;
29. Inability to swallow capsules or refractory nausea and vomiting, malabsorption, external bile diversion, or any significant small bowel resection that may interfere with the complete absorption of the study drug;
30. Researchers believe there are other situations that are not suitable for inclusion. For example, factors related to family or society may affect the safety of the subjects, or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-05-19 (Estimated); Primary Completion 2028-04-27 (Estimated); Study Completion 2028-04-27 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival | Evaluation of tumor burden based on RECIST criteria until first documented progress through study completion, an average of 6 weeks
  Time from treatment beginning until disease progression

SECONDARY OUTCOMES:
Objecitve response rate | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 6 weeks
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission
Disease control rate | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 6 weeks
  Proportion of patients who achieved a complete response, a partial response, or stable diseas
Duration of Response | Through study completion, an average of 3 weeks
  the time from the initial assessment of CR or PR for subjects with the best tumor efficacy to disease progression or death from any cause.
Overall Survival | From date of treatment beginning until the date of death from any cause, through study completion, an average of 3 weeks
  Time from treatment beginning until death from any cause
Incidence of Treatment-related adverse Events | Through study completion, an average of 3 weeks
Explore therapeutic efficacy biomarkers (including p-ERK levels, etc.) | Before the subjects start the study treatment

IPD SHARING:
Plan to Share IPD: No